CLINICAL TRIAL: NCT00291083
Title: Study of Manual Nipple Fluid Aspiration IN Post-Menopausal Women
Brief Title: Protocol for Postmenopausal Women at Increased Risk of Developing Breast Cancer
Status: Completed | Type: Observational
Sponsor: Carol Fabian, MD (Other)
Responsible Party: Sponsor-Investigator, Carol Fabian, MD, Professor, Director Breast Cancer Prevention Unit, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Other Study IDs: 8427
Record Dates: First submitted 2006-02-10; First posted 2006-02-13 (Estimated); Last update posted 2012-02-07 (Estimated); Status verified 2012-02

CONDITIONS: Breast Cancer
Keywords: NAF; nipple aspirate fluid; breast atypia; high risk for breast cancer; breast epithelial hyperplasia; Ki-67; hormones plus chemoprevention; chemoprevention
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To examine nipple aspirate fluid for secretions that may be identified as a high risk indicator for development of breast cancer, and compare those to serum analysis.

DETAILED DESCRIPTION:
To examine nipple aspirate fluid analysis in lactating women for local concentration of estrogen, prolactin, glucocorticoids, insulin, parity, prior lactation and age. NAF secretors have been reported to have modest increase in breast cancer risk compared to non-secretors . Estrogen levels have been found to be markedly higher in NAF samples than in the serum collected from the same women. Estradiol and estrone concentrations in premenopausal women are 10x and 20x greater in NAF samples than in serum and 50x and 35x greater in post-menopausal women not on HRT. It has been suggested that the disparity between serum and NAF levels may be due to local estrogen production via aromatase and sulfatase.

ELIGIBILITY:
Inclusion Criteria:

* women with high a high risk of breast cancer
* Older than 18

Exclusion Criteria:

* anticoagulants
* marked breast tenderness
* pregnant or within twelve months of breast feeding/childbirth

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Medical center
Sampling Method: Non-Probability Sample
Enrollment: 229 (Actual)
Dates: Start 2005-10; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol J Fabian, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States